CLINICAL TRIAL: NCT05367414
Title: The Effect of Aromatherapy Massage on Itching, Comfort, Skin pH Level, and Skin Moisture in Liver Diseases: Randomised Controlled Trial
Brief Title: Aromatherapy Massage for Itching Management in Liver Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amine Terzi (Other)
Responsible Party: Sponsor-Investigator, Amine Terzi, Asst. Prof., Artvin Coruh University
Organization: Artvin Coruh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Amine TERZİ
Record Dates: First submitted 2022-04-18; First posted 2022-05-10 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2022-05

CONDITIONS: Aromatherapy; Massage; Liver Diseases; Itching; pH Level; Skin Moisture
Keywords: aromatherapy; massage; liver Diseases; itching
MeSH Terms: conditions — Liver Diseases; Pruritus | interventions — almond oil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- aromatherapy (Experimental): In addition to routine medical treatment, massage with diluted tea tree oil was applied to the individuals in this group.
  Interventions: Other: aromatherapy massage (diluted tea tree oil)
- placebo (Placebo Comparator): Individuals in this group were provided massage with sweet almond oil in addition to routine medical treatment.
  Interventions: Other: aromatherapy massage (sweet almond oil)
- control (No Intervention): Individuals in this group received only routine medical treatment.

INTERVENTIONS:
Other: aromatherapy massage (diluted tea tree oil) — massage with diluted tea tree oil was applied
  Arms: aromatherapy
Other: aromatherapy massage (sweet almond oil) — massage with sweet almond oil was applied
  Arms: placebo

SUMMARY:
The aim of this study is to determine the effect of aromatherapy massage on itching, comfort, skin pH level and skin moisture in individuals with liver disease.

Research Hypotheses:

H1: Aromatherapy massage has an effect on the level of itching in individuals with itchy liver disease.

H2: Aromatherapy massage has an effect on the general comfort level in individuals with itchy liver disease, H3: Aromatherapy massage has an effect on skin pH level in individuals with itchy liver disease.

H4: Aromatherapy massage has an effect on skin moisture in individuals with itchy liver disease.

DETAILED DESCRIPTION:
This randomised controlled trial was conducted in order to examine study effect of aromatherapy massage on itching, comfort, skin pH level, and skin moisture among individuals with liver diseases

ELIGIBILITY:
Inclusion Criteria:

* patients who volunteered to participate in the study,
* with a diagnosis of chronic liver disease (liver cirrhosis (primary biliary cirrhosis, alcoholic, cardiac, post-necrotic, cryptogenic cirrhosis, Wilson's Cirrhosis, hemochromatosis), chronic viral hepatitis),
* had no cognitive impairment,
* were not included in the pre-application,
* could answer questions,
* itch score of above 3 (with Visual Analogue Scale).

Exclusion Criteria:

* patients are taking antipruritic treatment,
* have itchy skin disease before, ulcer, eczema, etc. in the area to be applied
* patients with dermatological problems, any swelling or signs of inflammation in the area ---to be treated, neuropathy or loss of sensation in the area to be treated
* patients with allergic to tea tree oil, perfume, or cosmetics,
* diagnosed with cancer

Ages: 37 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Itching | Day 1
  Itching was assessed with the 5D Itch Scale. The total score of the scale ranges from 5 to 25, with 5 points indicating the absence of itching and 25 points indicating the highest severity of itching.
Itching | Day 14
  Itching was assessed with the 5D Itch Scale. The total score of the scale ranges from 5 to 25, with 5 points indicating the absence of itching and 25 points indicating the highest severity of itching.
comfort | Day 1
  Comfort assessed with the General Comfort Scale. The score to be obtained from the scale varies between 48 and 192. 48 points indicating the low comfort level and 192 points indicating the high comfort level.
comfort | Day 2
  Comfort assessed with the General Comfort Scale.The score to be obtained from the scale varies between 48 and 192. 48 points indicating the low comfort level and 192 points indicating the high comfort level.
comfort | Day 14
  Comfort assessed with the General Comfort Scale. The score to be obtained from the scale varies between 48 and 192. 48 points indicating the low comfort level and 192 points indicating the high comfort level.
skin pH level | Day 1
  For pH level measurement, the F-74 G model skin pH measuring device manufactured by HORIBA Scientific and ISFET (Ion Sensitive Field Effect Transistor) 0040-10D model pH electrode produced by HORIBA Scientific were used.
skin pH level | Day 2
  For pH level measurement, the F-74 G model skin pH measuring device manufactured by HORIBA Scientific and ISFET (Ion Sensitive Field Effect Transistor) 0040-10D model pH electrode produced by HORIBA Scientific were used.
skin pH level | Day 14
  For pH level measurement, the F-74 G model skin pH measuring device manufactured by HORIBA Scientific and ISFET (Ion Sensitive Field Effect Transistor) 0040-10D model pH electrode produced by HORIBA Scientific were used.
skin moisture level | Day 1
  DMM brand skin moisture measuring device was used to measure skin moisture level.
skin moisture level | Day 2
  DMM brand skin moisture measuring device was used to measure skin moisture level.
skin moisture level | Day 14
  DMM brand skin moisture measuring device was used to measure skin moisture level.

CONTACTS AND LOCATIONS:
Overall Officials: Amine TERZI, PHD, Principal Investigator — Artvin Coruh University; Yasemin YILDIRIM, PHD, Study Director — Ege University; Fisun SENUZUN AYKAR, PHD, Study Chair — Izmir Tinaztepe University; Ulus Salih AKARCA, PHD, Study Chair — Ege University
Locations (1):
- Artvin Coruh University, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No